CLINICAL TRIAL: NCT05686278
Title: A Post-market Clinical Follow-up (PMCF) Study to Evaluate Clinical, Radiographic and Patient Reported Outcomes Following a Hip Hemiarthroplasty Surgery Using Corin Devices
Brief Title: Observational Study to Evaluate Long-Term Outcome in Hip Hemiarthroplasty
Status: Recruiting | Type: Observational
Sponsor: Corin (Industry)
Responsible Party: Sponsor
Other Study IDs: CSP2021-05-FR
Record Dates: First submitted 2023-01-06; First posted 2023-01-17 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Hip Fractures; Hip Hemiarthroplasty; Osteoarthritis, Hip; Avascular Necrosis of Hip; Femoral Neck Fractures
Keywords: Hemiarthroplasty; Acetabulum; Hip Fractures
MeSH Terms: conditions — Hip Fractures; Osteoarthritis, Hip; Femoral Neck Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hip hemiarthroplasty with BiPolar i and cemented stems (Meije or Oceane+): Subjects clinically suitable for a hip hemiarthroplasty surgery with Corin hip devices
  Interventions: Device: Bipolar i and cemented stem (Océane+ or Meije)

INTERVENTIONS:
Device: Bipolar i and cemented stem (Océane+ or Meije) — Hip hemiarthroplasty is a surgical procedure that involves replacing half of the hip joint

SUMMARY:
This PMCF study is designed to collect safety and efficacy data on hip hemiarthroplasty surgeries with Corin BiPolar-i shell and the Oceane+ or Meije Duo femoral stem up to 10 years.

DETAILED DESCRIPTION:
As part of the current clinical remediation work under the new Medical Device Regulation (MDR), limited data have been identified to support the hemiarthroplasty indication for some of Corin femoral stems. Therefore, this PMCF study has been implemented to collect safety and performance data on hip hemiarthroplasty surgeries with Corin BiPolar-i shell and the Oceane+ or Meije Duo femoral stem up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders.
2. Adult subjects.
3. Subjects clinically suitable for a hip hemiarthroplasty surgery with Corin hip devices based on physical examination, medical history and diagnosis such as: non-inflammatory degenerative joint disease including osteoarthritis and avascular necrosis in which the acetabulum does not require replacement, treatment of non-union, femoral neck and trochanteric fractures of the proximal femur, revision of failed partial hip replacements in which the acetabulum does not require replacement.
4. The subject is willing to comply with the required follow-up visits as per protocol.
5. The subject has signed a Patient Informed Consent Form (PICF), specific to this study, and approved by the local EC.

Exclusion Criteria:

1. Subjects with active infection or sepsis or osteomyelitis.
2. Subjects with unsuitable or insufficient bone support preventing proper fixation of the prosthesis.
3. Subject with marked bone loss or bone absorption.
4. Subject with metabolic disorders which may impair bone formation or bone quality.
5. Subjects under guardianship.
6. Subjects in the opinion of the Investigator/ investigative team who will be unable to comply with study procedures (Examples: recent psychotic or mania disorders, alcohol, drug or substance abusers) and/or those unable for any medical or other reason to comply with study procedures/visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects clinically suitable for a hip hemiarthroplasty surgery with Corin hip devices based on physical examination, medical history and diagnosis such as: non-inflammatory degenerative joint disease including osteoarthritis and avascular necrosis in which the acetabulum does not require replacement, treatment of non-union, femoral neck and trochanteric fractures of the proximal femur, revision of failed partial hip replacements in which the acetabulum does not require replacement.
Sampling Method: Non-Probability Sample
Enrollment: 368 (Estimated)
Dates: Start 2023-06-29 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2033-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation of safety of the study devices at 2 years after a hip hemiarthroplasty surgery. | 2 years
  Intraoperative and postoperative adverse events (hip, device or procedure related) will be recorded.

SECONDARY OUTCOMES:
Evaluation of mid-term and long-term safety of the study devices up to 10 years. | 10 years
  Intraoperative and postoperative adverse events (hip, device or procedure related) will be recorded.
Evaluation of study devices performance and benefit through patient's mobility from baseline to 10-year FU. | 10 years
  Parker Mobility Score
Evaluation of study devices performance and benefit through patient's quality of life from baseline to 10-year FU. | 10 years
  EQ5D-5L
Radiographic analysis to detect acetabular erosion | 2 years
  Acetabular erosion measured comparing immediate post-operative X-rays (baseline) to 2-year follow up and classified according to the criteria of Baker et al.
Radiographic analysis to detect femoral stem stability | 2 years
  Femoral stem stability measured on weight-bearing AP and lateral X-rays as rate of continuous, progressive and symptomatic periprosthetic radiolucent lines greater than 2mm using the zonal classification described by Gruen et al. from immediate postoperative (baseline) to 2-year follow up.
Radiographic analysis to detect bipolar head migration | 2 years
  Bipolar head migration measured comparing immediate post operative X Rays (baseline) to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Christophe HULET, MD, PhD, Study Chair — University Hospital, Caen
Locations (3):
- France (3):
  - Ch Amboise, Amboise
  - Polyclinique Henin Beaumont, Hénin-Beaumont
  - Hopital Saint Joseph, Paris